CLINICAL TRIAL: NCT01260545
Title: Phase I Study of CA-18C3 in Subjects With Advanced Hematologic Malignancies
Brief Title: Study of CA-18C3 in Subjects With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-PT015
Record Dates: First submitted 2010-12-10; First posted 2010-12-15 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — bermekimab

ARMS (1):
- Infusion (Experimental): A standard 3+3 design will be employed to determine maximum tolerated dose
  Interventions: Drug: CA-18C3

INTERVENTIONS:
Drug: CA-18C3 — 2.5 mg/kg, 3.75 mg/kg IV (in the vein) on Day 1 of each 14 day cycle until the subject is no longer benefiting clinically or unacceptable toxicity occurs.

SUMMARY:
The purpose of this study is to examine the safety and tolerability of CA-18C3 in subjects with hematologic malignancies, as well as look at the preliminary efficacy of IL-1alpha blockade.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age ≥ 18 years of age
* Subject must have a relapsed/refractory leukemia for which no standard therapies are anticipated to result in a durable remission. Subjects with previously treated high-risk myelodysplasia (MDS) (Intermediate 2 or high-risk by IPSS) and chronic myelomonocytic leukemia-2 (CMML-2 by WHO classification) are also candidates for this protocol. Relapsed/refractory leukemias include acute non-lymphocytic leukemia (AML) by WHO classification, acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), or chronic myelogenous leukemia (CML) in blast crisis. Subjects with myelofibrosis are also eligible. Untreated patients with above diagnoses considered unfit for standard therapy will also be eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
* Women of child bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative urine pregnancy test within 2 weeks prior to beginning treatment on this trial. Nursing subjects are excluded. Sexually active men must also use acceptable contraceptive methods for the duration of time on study. Pregnant and nursing subjects are excluded because the effects of CA-18C3 on a fetus or nursing child are unknown.
* In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for non-cytotoxic agents. If the subject is on hydroxyurea to control peripheral blood leukemic cell counts, the subject must be off hydroxyurea for at least ¬48 hours before initiation of treatment on this protocol. Persistent clinically significant toxicities from prior chemotherapy must not be greater than grade 1.
* Subjects must have the following clinical laboratory values (unless out of range values are considered to be the result of leukemic organ involvement):

  1. Serum creatinine ≤ 2.0 mg/dl.
  2. Total bilirubin ≤ 1.5x the upper limit of normal unless considered due to Gilbert's syndrome.
  3. Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) ≤ 3x the upper limit of normal unless considered due to organ leukemic involvement.
* Signed and dated institutional review board (IRB)-approved informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure.
* Subjects receiving any other standard or investigational treatment for their hematologic malignancy.
* Subjects who at the time of evaluation for participation in the study have evidence of active leukemic involvement in the brain or spinal cord (CNS).
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* Subjects immunocompromised due to a process unrelated to leukemic disease or treatment, including subjects known to be infected with human immunodeficiency virus (HIV)
* Subjects with detectable levels of endogenous antibodies to IL-1α at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04-30 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2012-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of CA-18C3, as well as the pharmakokinetic properties of CA-18C3 in study participants. | one year
  To determine the toxicities, including the dose limiting toxicity and maximum tolerated dose of CA-18C3 when administered intravenously at up to 3.75 mg/kg twice monthly in subjects with hematologic malignancies.
  To determine the pharmacokinetics (PK) of CA-18C3 following study drug administration

SECONDARY OUTCOMES:
Number of participants with disease progression, stable disease, partial response or complete response of their disease while receiving CA-18C3. | One year
  To observe the anti-tumor effects of CA-18C3, if any occur

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States